CLINICAL TRIAL: NCT03329079
Title: Engaging Rural Men With Mobile Technologies for Weight Loss: A Randomized Controlled Trial.
Brief Title: Engaging Rural Men With Mobile Technologies for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Northeast Nebraska Public Health Department (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0594-17-EP
Record Dates: First submitted 2017-10-18; First posted 2017-11-01 (Actual); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Weight Loss
Keywords: rural; men; community-based participatory research; weight loss; mobile applications; text messaging
MeSH Terms: conditions — Weight Loss; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Masking Description: The assessor will know which group assignment the subject has been given as is required for him to download the appropriate app and provide training on the technology to the subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Technology Plus (MT+) (Experimental): Experimental arm will receive a 3-month MT+ intervention using the premium mobile phone app version with social comparison group, behavior change text messaging, and daily self-weighing via Wi-Fi scale.
  Interventions: Behavioral: Mobile Technology Plus
- Mobile Technology (MT) (Active Comparator): Comparison group will receive the basic version of the mobile phone app only.
  Interventions: Behavioral: Mobile Technology

INTERVENTIONS:
Behavioral: Mobile Technology Plus — The intervention group MT+ will receive the premium-version mobile phone app with social comparison group, behavior change text messaging, and daily self-weighing via Wi-Fi scale.
  Other Names: MT+
  Arms: Mobile Technology Plus (MT+)
Behavioral: Mobile Technology — The comparison group MT will receive the basic-version mobile phone app only to self monitor eating, activity, and weight.
  Other Names: MT
  Arms: Mobile Technology (MT)

SUMMARY:
Overweight and obese men in rural Northeast Nebraska are an unrepresented, at-risk group exhibiting rising rates of cardiovascular disease, poor access to preventive care, and a rural milieu that contributes to their sedentary physical activity and unhealthy diet. This study proposes to use a pragmatic randomized controlled trial and community engaged research approaches to 1) determine the feasibility and acceptability of a commercially available, smart phone self-monitoring app (premium-version) plus text-based coaching and daily weighing via Wi-Fi scale intervention for achieving weight loss, 2) determine preliminary efficacy of this intervention group to a comparison group receiving only a self-monitoring app (basic-version) in achieving the outcomes of weight loss (kilogram) and improved dietary and physical activity behaviors (secondary) at 6 months post-baseline, and 3) determine quantitative and qualitative indicators of community capacity to support a contextually relevant weight loss intervention. Eighty men (ages 40-69) with body mass index of 28 or higher, randomly assigned (1:1 ratio) to intervention group or comparison group. Men will complete baseline assessments (weight, % body fat, body mass index height, blood pressure, health history, dietary intake, physical activity frequency/intensity) and receive orientation to the mobile technologies (app features, text messaging, Wi-Fi scale). Men will track their dietary intake, physical activity, and weight on the app for 12 weeks. After the 3-month intervention, post-measure assessments (weight, % body fat, BMI, dietary intake, PA frequency/intensity, technology usability surveys) will be collected at 3 and 6 months post-baseline. At 6 months post-baseline, two groups (n=8 each) of intervention completers will be purposively selected to share their perceptions of the intervention efficacy in an evaluative focus group. A community advisory board comprising local leaders within the men's social network, together with investigators and rural student nurses will guide community outreach efforts for study recruitment, implementation and evaluation. Study findings will be evaluated with the community to inform local dissemination, future intervention revision, and determination of community capacity for support of a larger clinical trial.

DETAILED DESCRIPTION:
Obesity is a major public health problem that disproportionately affects rural men and promotes the development of chronic conditions such as diabetes, cardiovascular disease, arthritis, and cancer. This study proposes to evaluate a mobile self-monitoring application (app) with Wi-Fi scale and text messaging intervention (MT+: mobile technology plus) for achieving weight loss in overweight and obese rural men. This proposal aligns with 1) Healthy People 2020's aim to eliminate health disparities by increasing physical activity and reducing obesity in adults; 2) the NIH's strategic plan to prioritize obesity reduction research among underserved rural populations; and, 3) the NINR's strategic focus on technology to promote health. Sixty nine percent of rural men in Nebraska are overweight or obese with increasing prevalence during midlife 40-59 (40%) and older (36%). Rural men are more likely to smoke, be obese, be physically inactive, and have shorter lifespans (2 years) than urban men. Rural men are also more likely to be uninsured/underinsured, less likely to engage in preventive health services, and report overall poorer health than urban men. Despite the burden of obesity, no self-monitoring mobile technology interventions targeting weight loss in rural, U.S. males exist, though the investigators preliminary study demonstrated rural men will use mobile technology for eating and activity self-monitoring. Studies show self-monitoring as one of the most effective behavior-change techniques for weight loss. MT+ provides an accessible means of real-time self-monitoring support for targeting lifestyle behaviors that lead to weight loss.

The investigators propose a pragmatic, randomized controlled trial (RCT) to examine the feasibility, acceptability, and preliminary efficacy of a MT+ intervention for weight loss in overweight and obese men in a practical, real-life rural environment. This 6-month pilot RCT includes a 3-month intervention with 6-month post-baseline follow-up. The intervention group (n=40) will receive a 3-month MT+ intervention using a commercially available, premium-version mobile phone app with social comparison group, behavior change text messaging, and daily self-weighing via Wi-Fi scale. The comparison group (n=40) will receive the basic-version mobile phone app only (MT). Primary efficacy outcome will be loss of body weight (kg & % body weight) at 3 and 6 months. Secondary outcomes will be improved diet and increased physical activity (PA). A multi-method formative evaluation of the intervention (student outreach, community advisory board (CAB), community capacity surveys, focus group, community dissemination) will occur across the study. Primary feasibility outcomes will include recruitment/retention rates and community resource development for program sustainment. The multi-modal feedback will help 1) facilitate recruitment of a hard-to-reach population, and 2) inform intervention feasibility and acceptability. These local insights may foster minimized attrition and improve future study outcomes. The specific aims of this study are:

Aim #1: Determine the feasibility and acceptability of a MT+ intervention for achieving weight loss in rural overweight and obese men. The aim will specifically address groups by the 1) participation rates including number of men recruited and randomized over a 6 month period. 2) retention rates, 3) feasibility, usability, satisfaction ratings, 4) adherence record of logging by men in the intervention group, and 5) evaluative focus group feedback.

Aim #2: Determine preliminary efficacy of a MT+ intervention to a comparison group receiving only a basic self-monitoring app (MT) in achieving 1) weight loss (primary), and 2) improved dietary and PA behavior (secondary) at 6 months post-baseline in rural men.

Aim #3: Determine quantitative and qualitative indicators of community capacity (resource mobilization, learning opportunities-skills development, partnership linkages, participatory decision-making, leadership) to support a relevant weight loss intervention for rural men.

Through a collaborative process guided by Community-Engaged Research (CEnR) approaches with a community-academic partnership involving UNMC students, community leaders, the investigators plan to create and disseminate local knowledge about obesity in rural men. Specifically, the investigators plan to 1) document the feasibility, acceptability, and preliminary efficacy of a weight loss intervention among rural men, a current gap in the NIH health disparities portfolio, 2) engage rural communities through student-informed outreach approaches and CAB partnership linkages to improve the efficacy of weight loss interventions for rural men, and 3) strengthen the research environment of the University of Nebraska Medical Center (UNMC) institution through providing opportunities for undergraduate and graduate students to conduct CEnR.

ELIGIBILITY:
Inclusion Criteria:

* Man age 40-69
* Reside in Northeast Nebraska
* BMI of 28 (kg/m2) or higher (BMI greater than 50 with clinician clearance, maximum weight 396 pounds)
* Smart phone owner with enabled text messaging
* Have an email account
* Answer "no" to all questions on the PAR-Q 17 health history assessment or are willing to get physician evaluation prior to enrolling
* Willing to share self-monitoring logs of eating, activity, and weight with investigative team.

Exclusion Criteria:

* Have recently lost 5% or more of body weight
* Are currently taking medications that cause or are influenced by weight loss
* Have used weight loss app in the past to lose weight
* Family member from same household is enrolled in this study
* Type I diabetes or Type II diabetes with insulin dependence

Ages: 40 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based upon self-representation of gender identity.
Enrollment: 80 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Berger, PhD, Study Director — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Norfolk, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Summary results will be shared with all identifiers removed at the completion of the study after all analyses have been finalized.

REFERENCES:
- [Background] Eisenhauer CM, Hageman PA, Rowland S, Becker BJ, Barnason SA, Pullen CH. Acceptability of mHealth Technology for Self-Monitoring Eating and Activity among Rural Men. Public Health Nurs. 2017 Mar;34(2):138-146. doi: 10.1111/phn.12297. Epub 2016 Oct 18. PMID 27757986
- [Background] Hageman PA, Pullen CH, Yoerger M. Physical Function and Health-Related Quality of Life in Overweight and Obese Rural Women Who Meet Physical Activity Recommendations. J Aging Phys Act. 2018 Jul 1;26(3):438-444. doi: 10.1123/japa.2017-0117. Epub 2018 Jun 13. PMID 28952857
- [Background] Hageman PA, Pullen CH, Hertzog M, Pozehl B, Eisenhauer C, Boeckner LS. Web-Based Interventions Alone or Supplemented with Peer-Led Support or Professional Email Counseling for Weight Loss and Weight Maintenance in Women from Rural Communities: Results of a Clinical Trial. J Obes. 2017;2017:1602627. doi: 10.1155/2017/1602627. Epub 2017 Apr 5. PMID 28480078
- [Background] Eisenhauer CM, Brito FA, Yoder AM, Kupzyk KA, Pullen CH, Salinas KE, Miller J, Hageman PA. Mobile technology intervention for weight loss in rural men: protocol for a pilot pragmatic randomised controlled trial. BMJ Open. 2020 Apr 14;10(4):e035089. doi: 10.1136/bmjopen-2019-035089. PMID 32295776
- [Background] Eisenhauer CM, Brito F, Kupzyk K, Yoder A, Almeida F, Beller RJ, Miller J, Hageman PA. Mobile health assisted self-monitoring is acceptable for supporting weight loss in rural men: a pragmatic randomized controlled feasibility trial. BMC Public Health. 2021 Aug 18;21(1):1568. doi: 10.1186/s12889-021-11618-7. PMID 34407782
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile Technology Plus (MT+) | Mobile Technology (MT)
Started | 40 | 40
Completed | 36 | 38
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Technology Plus (MT+) | Mobile Technology (MT) | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.06 (8.15) | 54.35 (9.10) | 54.20 (8.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 40 | 40 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 39 | 39 | 78
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 40 | 38 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Weight by Randomized Group
Description: Weight in kilograms (as measured on a Tanita brand digital scale, TBF-215 Tanita Corporation of America)
Time Frame: Observed means from baseline weight and at 6 months
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Mobile Technology Plus (MT+) | Mobile Technology (MT)
Number analyzed (Participants) | 36 | 38
kilograms | -7.03 (2.9) | -4.14 (5.85)

2. Secondary Outcome: Point Estimate and Variability of Outcome Measure for Fruit and Vegetable Intake
Description: daily fruit and vegetable servings (Brief Risk Factor Surveillance Survey written questionnaire- Fruit and vegetable dietary intake module (Reported total number of fruit and vegetable serving sizes per 24 hour period)
Time Frame: Observed means from baseline fruit and vegetable intake at 6 months
Measure: Mean (Standard Deviation); unit: servings per day
Arm/Group | Mobile Technology Plus (MT+) | Mobile Technology (MT)
Number analyzed (Participants) | 36 | 37
servings per day | 3.16 (1.67) | 3.09 (1.54)

3. Secondary Outcome: Point Estimate and Variability of Outcome Measure for Beverage Intake Quality
Description: sugar-sweetened total beverage energy intake (Sugar Sweetened beverage intake questionnaire (BEV-Q15) Reported total number of fluid ounces consumed per 24 hour period)
Time Frame: Observed means from baseline beverage intake and at 6 months
Measure: Mean (Standard Deviation); unit: fluid ounces per day
Arm/Group | Mobile Technology Plus (MT+) | Mobile Technology (MT)
Number analyzed (Participants) | 36 | 38
fluid ounces per day | 4.34 (6.44) | 10.58 (17.01)

4. Secondary Outcome: Point Estimate and Variability of Outcome Measure for Physical Activity
Description: total steps taken in 24 hour period (Automated app report of total steps measured via gyroscope on smart phone- total step count range 0-10,000 steps (higher step value represents desired outcome of 10,000 steps per day)
Time Frame: Observed means from baseline overall physical activity and at 6 months
Measure: Mean (Standard Deviation); unit: Activity steps as measured by phone app
Arm/Group | Mobile Technology Plus (MT+) | Mobile Technology (MT)
Number analyzed (Participants) | 28 | 25
Activity steps as measured by phone app | 6874.64 (4650.58) | 5359.50 (2995.44)

ADVERSE EVENTS:
Time Frame: 1 year, 5 months
Arm/Group | Mobile Technology Plus (MT+) | Mobile Technology (MT)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT03329079/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT03329079/ICF_001.pdf